CLINICAL TRIAL: NCT05861518
Title: Effect of Hypnosis on Pain, Anxiety, and Quality of Life in Female Patients With Fibromyalgia: A Randomized Study
Brief Title: The Effect of Hypnosis in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Seyda Efsun Ozgunay, Asocc Prof, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-KAEK-25 2019/12-15
Record Dates: First submitted 2023-04-12; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Analgesia; Anxiety; Depression; Hypnosis
Keywords: fibromyalgia; hypnosis; depression; anxiety; analgesia
MeSH Terms: conditions — Agnosia; Anxiety Disorders; Depression; Fibromyalgia | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: collecting data and continuing treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): .Participants, who had been receiving treatment for FMS for at least six months at the physical therapy and rehabilitation outpatient clinic .Participants continued their current drug treatment. In the hypnosis group, the patients were given 3 hypnosis sessions once a week. in groups of 3, each standardized for approximately 30 minutes.
  Interventions: Behavioral: Hypnosis
- Group 2 (No Intervention): .Participants, who had been receiving treatment for FMS for at least six months at the physical therapy and rehabilitation outpatient clinic .Participants continued their current drug treatment.

INTERVENTIONS:
Behavioral: Hypnosis — In the hypnosis group, patients were given hypnosis sessions of approximately 30 minutes each, in groups of three, once a week. In this way, session standardization was achieved. Arm catalepsy was suggested in all patients. The first session was used as hypnosis induction, progressive muscular relaxation and introduction to hypnosis. In the second session, in addition to the first session, self-hypnosis training was given. The second session was applied as the same 3rd session. In these patients, in addition to analgesia suggestions, the feeling of worthlessness was especially studied with the recommendation of a psychiatrist.
  Arms: Group 1

SUMMARY:
Fibromyalgia syndrome (FMS) is a chronic disease characterized by widespread pain of unknown origin, fatigue, sleep disturbances, and cognitive problems. In the treatment of FMS, it is known that pharmacological therapy reduces fatigue as well as pain, increases functionality, and has positive effects on general well-being. In functional magnetic resonance imaging (fMRI) studies, suggestion following hypnotic induction has been reported to be better at pain control in patients with FMS. Self-hypnosis is a technique performed by the patient himself. The patients were randomly divided into two groups using the closed envelope technique as Group 1: Hypnosis and Group 2: Control. Patients who had communication problems, had other rheumatological diseases, had major medical disease and received treatment, had neurological and/or central nervous system disease, had been using antipsychotic medication, had been treated with psychotherapy for the last three months, and did not want to participate in the study were excluded from the study. Demographic characteristics of the participants and fibromyalgia effect beck depression and anxiety scale, Nottingham health profile and Visual Analogue Scale (VAS) were applied and the results were recorded. At the end of the 6th month, all scales and patient controls were made and re-evaluated.

In this study, we aimed to evaluate the effects of controlled, standardized adjuvant hypnosis on pain, depression, anxiety, aerobic exercise practices, quality of life, and disease impact score in patients with FMS who had been under treatment for at least six months.

DETAILED DESCRIPTION:
In the hypnosis group, the patients received hypnosis sessions of approximately 30 minutes each, in groups of three, once a week. During the first meeting with the hypnotist, information on hypnosis was given, and the method to be used was explained. Hypnosis was performed by a single practitioner. The first session included hypnosis induction, progressive muscular relaxation, and introduction to hypnosis. In the second session, in addition to the brief repetition of the first session, self-hypnosis training was given. The third session was applied the same way as the second session. While the hypnosis session focused on relaxation and pain, aerobic exercises were also suggested as a regular practice. In addition, self-hypnosis practices were suggested at least three days a week.The results of the scales administered to the participants at baseline were recorded, and these evaluations were repeated at the end of the sixth month. During the six-month period, all patients continued their current medical therapy.

This is a randomized study showing the effects of standardized hypnosis and self-hypnosis as adjuvant on VAS, FIQ, depression, anxiety and NHL in patients with FMS.

ELIGIBILITY:
Inclusion Criteria:

* Female
* FMS patients
* 35 to 65 years
* receiving treatment for FMS for at least six months

Exclusion Criteria:

* Patients with communication problems
* other rheumatological diseases
* major another medical diseases
* neurological and/or central nervous system diseases
* severe mental illnesses
* antipsychotic medication use

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 35-65
Enrollment: 50 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
VAS | the changes in scale scores from baseline to sixth month
  Visual Analogue Scale (VAS) was used to determine the severity of pain and fatigue of the patients.(from 0 better, 10 the worse) on a 10 cm line in VAS
depression scale | the changes in scale scores from baseline to sixth month
  Beck depresion scale (BDI): BDI measures physical, emotional, cognitive, and motivational symptoms seen in depression. It is a self-assessment scale that includes 21 symptom categories. The highest score that can be obtained is 63, with a higher total score indicating a greater severity of depression.
anxiety | the changes in scale scores from baseline to sixth month
  Beck anxiety scale (BAI): BAI measures the frequency of anxiety symptoms experienced by an individual. It is a Likert-type self-assessment scale consisting of 21 items, each scored between 0 and 3. A high total score indicates a high level of anxiety experienced by the person.
Fibromyalgia | the changes in scale scores from baseline to sixth month
  Fibromyalgia Impact Questionnaire (FIQ): Except for the well-being property, low scores indicate recovery or less affliction. The maximum possible score on each subscale is 10, and the maximum total score that can be obtained is 100.
Health Profile | the changes in scale scores from baseline to sixth month
  Nottingham Health Profile (NHP): It contains a total of 38 questions in six areas: pain, physical abilities, energy level, sleep, social isolation, and emotional reaction. The response options for each item are "yes" and "no". Each subarea is scored between 0 and 100, with 0 indicating good health and 100 representing poor health

SECONDARY OUTCOMES:
exercise | at six month later
  the patient continues to exercise at the recommended frequency (3 times a week)

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa yüksek ihtisas EAH, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Study protocol can be share.
Supporting Information: Study Protocol
Time Frame: One year
Access Criteria: For academic studies